CLINICAL TRIAL: NCT02257424
Title: BRAF, Autophagy and MEK Inhibition in Metastatic Melanoma: A Phase I/II Open-Label Trial of Dabrafenib, Trametinib and Hydroxychloroquine in Patients With Advanced BRAF Mutant Melanoma
Brief Title: Dabrafenib, Trametinib and Hydroxychloroquine in Patients With Advanced BRAF Mutant Melanoma
Acronym: BAMM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 02614
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Advanced BRAF Mutant Melanoma
MeSH Terms: interventions — trametinib; Hydroxychloroquine; dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase 1/2 (Other)
  Interventions: Drug: Trametinib 2 mg daily; Drug: hydroxychloroquine (HCQ); Drug: dabrafenib 150 mg orally twice a day

INTERVENTIONS:
Drug: Trametinib 2 mg daily
Drug: hydroxychloroquine (HCQ) — hydroxychloroquine (HCQ) is 600 mg orally every 12 hours
Drug: dabrafenib 150 mg orally twice a day

SUMMARY:
The primary purpose of this study is to determine the maximum tolerated dose (MTD) and preliminary safety of hydroxychloroquine (HCQ) when administered in conjunction with oral dabrafenib and trametinib (D+T) in patients with advanced BRAF mutant melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age.
* Patients must have histologically confirmed melanoma unresectable Stage III or Stage IV positive for BRAF V600E, V600K, V600R or V600D by a CLIA approved assay.
* Patients must have an ECOG performance status of 0 or 1.
* Patients must have adequate baseline organ function as determined by table 2.

Table 2. Definitions for adequate baseline organ function

Laboratory Values

Hematologic:

* ANC (absolute neutrophil count) ≥1.2 × 109/L
* Hemoglobin ≥ 9 g/dL
* Platelet count ≥100 x 109/L
* PT/INR and PTT ≤ 1.3 x ULN (PT = prothrombin time; INR = international normalized ratio; PTT = partial thromboplastin time; ULN = upper limit of normal)

Hepatic

* Total bilirubin ≤ 1.5 x ULN
* AST (aspartate aminotransferase) and ALT (alanine transaminase) ≤ 2.5 x ULN

Renal -- Serum creatinine ≤ 1.5 mg/dL

Cardiac

-- Left Ventricular Ejection fraction (LVEF) ≥ LLN (lower limit of normal) by ECHO

Subjects receiving anticoagulation treatment may be allowed to participate with INR established within the therapeutic range prior to randomization.

If serum creatinine is > 1.5 mg/dL, calculate creatinine clearance using standard Cockcroft-Gault formula. Creatinine clearance must be ≥ 50 mL/min to be eligible.

Except subjects with known Gilbert's syndrome. ECHO scans must be used throughout the study when indicated

* Patients must be able to provide written informed consent.
* Negative serum pregnancy test within 7 days prior to commencement of dosing in premenopausal women. Women of non-childbearing potential may be included without serum pregnancy test if they are either surgically sterile or have been postmenopausal for ≥ 1 year. Women must use an effective method of contraception from 14 days prior to randomization, throughout the treatment period, and for at least 6 months after the last dose of study treatment as directed by their physician. Effective methods of contraception are defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly (for example implants, injectables, or intra-uterine devices). At the discretion of the investigator, acceptable methods of contraception may include total abstinence in cases where the lifestyle of the patient ensures compliance. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.) Hormonal-based methods (e.g., oral contraceptives) are NOT permitted as contraception due to potential drug-drug interactions with dabrafenib.
* Patients with brain metastases treated with whole brain radiation that have been stable for 2 months are eligible; patients with brain metastases treated with gamma knife or surgery are allowed to participate after 2 weeks have elapsed since their procedure. Subjects are excluded if they have leptomeningeal or metastases causing spinal cord compression that are symptomatic or untreated or not stable for ≥3 months (must be documented by imaging) or requiring corticosteroids. Subjects on a stable dose of corticosteroids >1 month or who have been off of corticosteroids for at least 1 week can be enrolled with approval of the medical monitor
* Any number and type of prior anticancer therapies are allowed except BRAF or MEK inhibitors .
* Patients must have discontinued active immunotherapy (IL-2, interferon, CTLA-4, etc.) or chemotherapy at least 4 weeks prior to entering the study and oral targeted therapy at least 2 weeks prior to entering the study. Patients must not receive any other investigational anticancer therapy during the period on study or the four weeks prior to entry.
* All prior anti-cancer treatment-related toxicities (except alopecia and laboratory values as listed in Eligibility Criteria #4) must be Grade 1 according to the Common Terminology Criteria for Adverse Events version 4 (CTCAE version 4.03, 2009) at the time of starting treatment. Patients that are asymptomatic on low dose maintenance hormone replacement delivered at a stable dose for prior toxicities are eligible.
* Patient much have measurable disease as defined by RECIST 1.1.
* Patients must be able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.

Exclusion Criteria:

* Patients with known serious concurrent infection or medical illness, including psychiatric disorders, which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety.
* Patients who are pregnant or breast-feeding.
* Patients receiving concurrent therapy for their tumor (i.e. chemotherapeutics or investigational agents).
* Patients who are known to be experiencing an objective partial response to immunotherapy at the time of study enrollment
* History of malignancy other than disease under study within 3 years of study enrollment with exceptions below:

Exception: Subjects with a history of completely resected non-melanoma skin cancer, or subjects with indolent second malignancies are eligible

* History of malignancy with confirmed activating RAS mutation at any time. Note: Prospective RAS testing is not required. However, if the results of previous RAS testing are known, they must be used in assessing eligibility.
* History of interstitial lung disease or chronic pneumonitis
* Due to risk of disease exacerbation patients with porphyria or psoriasis are ineligible unless the disease is well controlled and they are under the care of a specialist for the disorder who agrees to monitor the patient for exacerbations.
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study drug, or excipients or to dimethyl sulfoxide (DMSO).
* Patients receiving cytochrome P450 enzyme-inducing anticonvulsant drugs (EIADs) (i.e. phenytoin, carbamazepine, Phenobarbital, primidone or oxcarbazepine) within 4 weeks of the start of the study treatment
* Current use of a prohibited medication as described in Section 6.3.8 of the protocol for Potential for Drug-Drug Interaction: apply moisturizing creams frequently, topical keratolytics (e.g. urea 20-40 % cream, salicylic acid 6%, tazarotene 0.1% cream, fluorouracil 5% cream), clobetasol propionate 0.05% ointment for erythematous areas, topical lidocaine 2%, and / or systemic pain medication such as nonsteroidal anti-inflammatory drugs, codeine, and pregabalin for pain.
* Known Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (subjects with laboratory evidence of cleared HBV and/or HCV will be permitted
* Patients with a previously documented retinal vein occlusion.
* History or evidence of increased cardiovascular risk including any of the following
* Left ventricular ejection fraction (LVEF) < institutional lower limit of normal.
* A QT interval corrected for heart rate using the Bazett's formula ≥ 480 msec;
* Current clinically significant uncontrolled arrhythmias. Exception: Subjects with controlled atrial fibrillation for >30 days prior to randomization are eligible.
* History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization.
* Current ≥ Class II congestive heart failure as defined by New York Heart Association
* Patients with intra-cardiac defibrillators
* Abnormal cardiac valve morphology (≥grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Phase 1: To determine the maximum tolerated dose | 5 weeks
  Phase 1: Maximum tolerated dose (MTD) = a) the dose producing Dose Limiting Toxicity (DLT) in 2/6 patients, or b) the dose level below the dose which produced DLT in ≥ 2/3 patients, or in ≥ 3/6 patients
Phase 2: To assess the clinical efficacy of HCQ+D+T by 1 year PFS rate. | 1 year
  Phase 2: Progression free survival (PFS) is defined as the duration of time from start of treatment to time of first progression, death due to any cause or last patient contact alive and progression-free

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Amaravadi, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (4):
- United States (4):
  - Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Amaravadi RK. Clinical trial results show promise of targeting autophagy BRAF mutant melanoma. Autophagy. 2022 Jun;18(6):1470-1471. doi: 10.1080/15548627.2022.2038899. Epub 2022 Feb 13. PMID 35156519